CLINICAL TRIAL: NCT04872283
Title: Prospective Randomized Study Evaluating the Effect of Postoperative Ketorolac on Bone Healing and Opioid Consumption After First Metatarsophalangeal Joint Fusion
Brief Title: Effect of Postoperative Ketorolac on Bone Healing After Joint Fusion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JONE19D.372
Record Dates: First submitted 2021-05-03; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Ketorolac; Joint Fusion
MeSH Terms: conditions — Ankylosis | interventions — Gene Fusion; Ketorolac; oxycodone-acetaminophen; Aspirin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded at enrollment and first made aware to which intervention they were randomized when receiving their postoperative pain medication at outside pharmacies
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketorolac administration (Active Comparator): Participants who have surgery for great toe (1st metatarsophalangeal joint) fusion will receive 30 mg of IV ketorolac during surgery as well as 20 mg ketorolac pills to take after surgery for pain
  Interventions: Procedure: great toe (1st metatarsophalangeal joint) fusion; Drug: IV Ketorolac; Drug: Ketorolac Pill; Drug: 5/325mg Oxycodone-Acetaminophen; Drug: Aspirin 81Mg Ec Tab
- No Ketorolac administration (Active Comparator): Participants who have surgery for great toe (1st metatarsophalangeal joint) fusion will receive the standard treatment of 30 tablets of oxycodone-acetaminophen to take as needed for pain
  Interventions: Procedure: great toe (1st metatarsophalangeal joint) fusion; Drug: 5/325mg Oxycodone-Acetaminophen; Drug: Aspirin 81Mg Ec Tab

INTERVENTIONS:
Procedure: great toe (1st metatarsophalangeal joint) fusion — Great Toe joint fusion surgery
Drug: IV Ketorolac — Participants will receive 30mg of intravenous (IV) ketorolac will be given during surgery
  Arms: Ketorolac administration
Drug: Ketorolac Pill — Participants will receive 20 tablets of 10mg ketorolac, with instructions to take 1 tablet orally every 6 hours for pain
  Arms: Ketorolac administration
Drug: 5/325mg Oxycodone-Acetaminophen — Participants will receive 30 tablets of 5/325mg oxycodone-acetaminophen with instructions to take 1 or 2 tablets by mouth every 4 to 6 hours as needed for pain
Drug: Aspirin 81Mg Ec Tab — Participants will receive 81 mg aspirin twice daily as a preventive measure against deep venous thrombosis (DVT)

SUMMARY:
In the midst of the opioid crisis, the use of non-narcotic pain medication has garnered increased interest, particularly in the field of orthopaedic surgery, where narcotic medications are routinely prescribed postoperatively. Nonsteroidal anti-inflammatory drugs (NSAIDs) have the potential to serve as an adjunct analgesic, but many orthopaedic surgeons have viewed NSAIDs with hesitancy because of evidence that they can lead to delayed bone healing.

When evaluating bone healing across different NSAID formulas, ketorolac was found to cause no delay and lead to better union rates when compared to controls and other NSAIDs, respectively. Previous studies in the orthopaedic spine and trauma literature have suggested a detrimental effect of NSAIDs, specifically ketorolac, with regards to bone healing, while others have reported no delay in healing. A recent study from our institution found no detrimental effects on the healing of ankle fractures with the use of ketorolac in the immediate postoperative period. Additionally, the use of ketorolac was associated with less reliance on narcotic pain medications.

The purpose of this prospective randomized study is to evaluate the use of ketorolac on postoperative pain, opioid requirements, patient satisfaction, complication/reoperation rates, and delayed and/or nonunion rates in patients undergoing fusion of their first metatarsophalangeal joint (1st MTPJ) for treatment of end-stage arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 undergoing outpatient primary 1st MTPJ fusion by a fellowship-trained foot and ankle orthopaedic surgeon at the Rothman Orthopaedic Institute

Exclusion Criteria:

* Patients undergoing revision 1st MTPJ fusion;
* Patients with any allergies to any study medication;
* Patients with documented chronic narcotic use;
* Patients with renal insufficiency, as defined by history and preoperative creatinine level (Cr ≥ 2.1 mg/dl);
* Patients who are pregnant;
* Patients undergoing inpatient procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 7 days
  Participants will be asked to complete the Visual Analog Scale for Pain Survey to measure postoperative pain
Satisfaction with pain management | 7 days
  This will be measured using the 6-point Likert scale (very dissatisfied, dissatisfied, slightly dissatisfied, slightly satisfied, satisfied, very satisfied)
Participant Perception of Pain | 7 days
  This will be measured using a 5-point Likert scale (never, almost never, often, almost always, always)

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States